CLINICAL TRIAL: NCT07071597
Title: The Selection of Initial Treatment Regimens for Adolescent Nephrotic Syndrome: A Multicenter Real-World Study.
Brief Title: The Selection of Initial Treatment Regimens for Adolescent Nephrotic Syndrome.
Status: Active, not recruiting | Type: Observational
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Yajing Xun, Principal Investigator, Nanjing Children's Hospital
Other Study IDs: 202412043-1
Record Dates: First submitted 2025-06-29; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Nephrotic Syndrome; Adolescent; Biopsy
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treatment Group: At the initial diagnosis, treatment is initiated with corticosteroids or immunosuppressive agents.
- Renal Biopsy Group: At the initial diagnosis, renal biopsy is performed first to clarify the renal pathology, and then targeted medication is used.
  Interventions: Procedure: Renal Biopsy

INTERVENTIONS:
Procedure: Renal Biopsy — Renal biopsy is performed to clarify the renal pathology.
  Groups: Renal Biopsy Group

SUMMARY:
Given that the treatment strategy for adolescent PNS has a significant impact on growth and development, but there are few cases and a lack of clinical research, this study plans to collaborate with several domestic top-tier children's nephrology centers to conduct a retrospective real-world study of adolescent PNS. The aim is to understand the current diagnosis and treatment status of adolescent PNS and compare the advantages and disadvantages of various therapies, in order to provide a more scientific, rational, and effective treatment plan for adolescent PNS.

DETAILED DESCRIPTION:
Pediatric kidney disease, especially primary nephrotic syndrome (PNS), is a common urinary system disease in pediatric clinical practice. The core pathophysiological process of nephrotic syndrome involves damage to the glomerular filtration membrane, resulting in massive proteinuria and subsequent hypoproteinemia, hyperlipidemia, and edema. PNS in children is more prevalent in the preschool age group, with minimal change disease (MCD) accounting for approximately 77.1% of pathological types. MCD is sensitive to corticosteroids, and the traditional initial treatment regimen is standard-dose corticosteroid induction therapy. In foreign countries, the pathological types of PNS in adolescents are mainly MCD and focal segmental glomerulosclerosis (FSGS). In mainland China, the proportion of mesangial proliferative glomerulonephritis (MsPGN) is increasing, but MCD remains the main pathological type. Currently, there is no consensus among guidelines from various countries on whether to perform renal biopsy and the indications for it in adolescent PNS. The Chinese pediatric PNS evidence-based guideline does not specify the age factor for renal biopsy. In the treatment protocol debate of the International Pediatric Nephrology Association (IPNA), some scholars advocate corticosteroid treatment first, while others believe that renal biopsy first can reduce steroid exposure and its side effects. However, there is still a lack of large-scale clinical data for comparison. Given that the treatment strategy for adolescent PNS has a significant impact on growth and development, but there are few cases and a lack of clinical research, this study plans to collaborate with several domestic top-tier children's nephrology centers to conduct a retrospective real-world study of adolescent PNS. The aim is to understand the current diagnosis and treatment status of adolescent PNS and compare the advantages and disadvantages of various therapies, in order to provide a more scientific, rational, and effective treatment plan for adolescent PNS.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis met the criteria for PNS from January 2014 to December 2023 (①Nephrotic-range proteinuria: 24-h urine protein ≥50 mg/kg or morning urine protein/creatinine (mg/mg) ≥2.0, three consecutive morning urine protein tests (＋＋＋) to (＋＋＋＋) within 1 week. ②Hypoproteinemia: serum albumin <25 g/L. ③Hyperlipidemia: serum cholesterol >5.7 mmol/L. ④Edema to varying degrees. Among the above four criteria, 1 and 2 are essential for diagnosis.);
2. Regular follow-up for at least 1 year;
3. Compliance with the requirements of the revised Helsinki Declaration of 2013, with informed consent obtained from patients and their families.

Exclusion Criteria:

1. Nephrotic syndrome secondary to other diseases;
2. Patients requiring dialysis or after kidney transplantation;
3. Presence of genetic defects or hereditary metabolic diseases;
4. Concurrent with severe primary diseases such as cardiovascular, liver, brain, hematopoietic system diseases, or mental disorders;
5. Incomplete clinical data.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Clinical data of PNS patients aged 10-18 years who met the diagnostic criteria for pediatric PNS established by the Pediatric Nephrology Group of the Chinese Medical Association in 2016, from multiple medical institutions over the past decade.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The number of relapses of proteinuria | From the start of treatment to 1 year and 2 years.
  The total number of proteinuria relapses in patients within 2 years of treatment is counted.
A 50% decline in kidney function | At 6 months, 1 year, and 2 years of treatment.
  Calculate the proportion of patients with a greater than 50% decline in kidney function at 6 months, 1 year, and 2 years of treatment.
Relapse-free rate of proteinuria after treatment | At 3 months, 6 months, 1 year, and 2 years after treatment initiation.
  The proportion of participants who remain free of proteinuria relapse after initial treatment, assessed by urine analysis and clinical evaluation.
Incidence of steroid resistance after treatment | At 4 weeks after treatment initiation.
  The proportion of participants who do not achieve remission with standard steroid therapy, assessed clinically and by laboratory evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Ruochen Che, Principal Investigator — Nanjing Children's Hospital
Locations (1):
- NanjingCH, Nanjing, China

IPD SHARING:
Plan to Share IPD: No